CLINICAL TRIAL: NCT06801327
Title: Comparison Between Different Respiratory Physiotherapy Techniques in Patients With Bronchiectasis. Conventional Therapy Versus Simeox: a Single-center, Randomized, Controlled, Cross-over Study
Brief Title: Comparison Between Conventional Respiratory Physiotherapy and the Simeox Device in Patients With Bronchiectasis
Acronym: FISIOBRONCHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FISIOBRONCHI
Record Dates: First submitted 2024-11-28; First posted 2025-01-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis Adult
Keywords: Bronchiectasis; Respiratory physioterapy; Simeox; Conventional respiratory physioterapy
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, open-label, 2x2 randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): Patients randomized to Group A will undergo the first treatment with conventional respiratory physiotherapy techniques (usually with Acapella, PEEP bottle, PEP mask, according to the standard clinical-assistance practice at our clinic and they will switch to Simeox for the second treatment
  Interventions: Device: Simeox
- Arm B (Other): Patients randomized to Group B will undergo the first treatment with Simeox, and they will switch to conventional respiratory physiotherapy techniques (usually with Acapella, PEEP bottle, PEP mask, according to the standard clinical-assistance practice at our clinicfor the second treatment
  Interventions: Device: Simeox

INTERVENTIONS:
Device: Simeox — The Investigators chose to evaluate this device for respiratory physiotherapy in our patients because it is the only one that offers innovative technology, as, unlike other commercially available devices, it does not require the patient to perform forced breathing. Instead, the patient can exhale calmly at tidal volume. This is expected to reduce the patient's effort and improve compliance with treatment. Furthermore, the vibratory signal with small, rapid, and sequential depressions within the airways could be more effective in mobilizing mucus from the airways, preventing collapse.

SUMMARY:
Physiotherapy is a key treatment for patients with bronchiectasis. An evaluation of the parameters indicative of respiratory health in patients treated with two different respiratory physiotherapy techniques (conventional versus Simeox®) would be very useful in choosing physiotherapy treatments for bronchiectasis patients. A systematic review of the literature shows that there are no published studies evaluating the effectiveness of respiratory physiotherapy by analyzing the variation in resistance measured using the forced oscillation technique (FOT) in patients with bronchiectasis. The results of this study would add to those that have examined different physiotherapy techniques and could therefore contribute to the choice of the most appropriate technique for this category of patients.

The trial is being conducted to answer the question: "How do respiratory parameters vary during treatment with two different respiratory physiotherapy techniques: conventional respiratory physiotherapy or that performed using the Simeox device?" Secondary objectives include the measurement of various functional parameters, such as vital signs (heart rate, respiratory rate, blood oxygenation, blood pressure values) and spirometry values (FEV1, FVC, TLC). The onset of adverse events, the degree of patient tolerance and relief, and respiratory health will also be assessed through the administration of various questionnaires commonly used in clinical practice. Additionally, changes in the quantity of sputum produced will be measured.

DETAILED DESCRIPTION:
Single-center, prospective, open-label, 2x2 randomized crossover study. It is planned to consecutively enroll all outpatient patients who attend the bronchiectasis clinic of the Pneumology and Respiratory Intensive Care Unit of the IRCCS, University Hospital of Bologna, Policlinico S. Orsola. The study has a 2x2 crossover design for superiority. Each enrolled patient will undergo two treatment periods, each lasting 4 weeks. Patients randomized to Group A will undergo the first treatment with conventional respiratory physiotherapy techniques (usually with Acapella, PEEP bottle, PEP mask, according to current clinical-assistance practice at our clinic), while patients randomized to Group B will start treatment with the Simeox® device.

At the end of the first 4 weeks, the treatment will be interrupted, and a 1-week wash-out period will be observed. Based on what is commonly observed in clinical practice, it is believed that 1 week of wash-out is adequate time for mucus to re-accumulate in the airways and restore the baseline conditions necessary for the crossover, while also avoiding the risk of adverse events due to mucus accumulation. At the end of the wash-out week, the second phase of the study will begin, also lasting 4 weeks, with a treatment switch: Group A patients will use the Simeox® device, and Group B patients will undergo conventional respiratory physiotherapy.

Randomization will be conducted with a 1:1 ratio without stratification by the statisticians of the Research and Innovation Unit of the IRCCS AOUBO using statistical software. The randomization list will be entered into the study's eCRF, created with REDCap, and will be consulted by the investigators at each new enrollment. Treatment arm assignment will be performed at V1.

If the enrolled patients are already undergoing respiratory physiotherapy, they will be subjected to a 1-week wash-out period before starting the study, during which respiratory physiotherapy will be suspended. The Investigators will not include patients with cystic fibrosis (CF) in the study, as the production of bronchial secretions in this group of patients is substantial. In patients with bronchiectasis not due to CF, however, secretion production is generally much more modest, and, as done in other studies, a short wash-out period does not significantly increase risks for these patients. For greater caution, the study will only be proposed to patients in a stable phase (absence of ongoing exacerbations) and with sputum production < 200 mL/day (comparable to 1 plastic cup). These are the criteria by which, in clinical judgment, "non-strongly secretive" patients are identified. During the wash-out period, patients will be invited to contact us immediately if sputum production exceeds 200 mL/day, in which case the investigators will exclude the patient from the study and arrange a short-term visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of bronchiectasis not due to cystic fibrosis who are not hospitalized.
* Age ≥ 18 years.
* Evidence of bronchiectasis in at least one lung lobe from a chest CT scan performed within the 10 years prior to enrollment.
* Absence of exacerbations in the 28 days preceding enrollment.
* Sputum producers with volumes less than or equal to 200 mL/day.
* Under treatment with optimized standard therapy for bronchiectasis that has been stable for at least one year, with no changes in the 28 days prior to enrollment.
* Eligible for and/or already undergoing respiratory physiotherapy.
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of COPD or bronchial asthma interpreted as primary and predominant diseases compared to bronchiectasis.
* Presence of tracheostomy.
* History of significant hemoptysis (≥300 mL of blood) or requiring embolization or blood transfusions in the 4 weeks preceding enrollment.
* Hemodynamic instability (mean arterial pressure < 65 mmHg, heart rate > 110 bpm).
* Undrained pneumothorax (evident on chest X-ray, deemed not worthy of pleural drainage according to standard clinical-assistance pathways and thus subjected to follow-up).
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of airway resistance | V1 (Baseline,) Visit 2 (Day 7), Visit 3 (Week 5), Visit 4 (Week 6), Visit 5 (Week 10)
  Airway resistance R5 and R20, measured in cmH2O/L/sec, using Forced Oscillometry Technique (FOT)

SECONDARY OUTCOMES:
Evaluation of Respiratory Rate | V1 (baseline), V3 (week 5), V5 (week 10)
  RR: Breath/Minutes
Evaluation of blood oxygen | At visits V1 (baseline), V3 (week 5), V5 (week 10)
  SpO2 (%)
Evaluation of hearth rate | At visits V1 (baseline), V3 (week 5), V5 (week 10)
  HR (bpm)
Evaluation of blood pressure | At visits V1 (baseline), V3 (week 5), V5 (week 10)
  Diastolic BP (mmHg) and Sistolic BP (mmHg)
Evaluation of spirometric values. | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  FEV1 (L), FVC (L), TLC (L) measured by Spirometry.
Evaluation of Six-minute walk test (6MWT) | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  Distance covered and vital parameters such as SpO2, heart rate, and respiratory rate at the beginning, at the end, and after recovery from exercise measured by pulse oximeter and calculation of distance walked.
Safety | V1 (Baseline,) Visit 2 (Day 7), Visit 3 (Week 5), Visit 4 (Week 6), Visit 5 (Week 10)
  Assessed in terms of the development of side effects and their severity. Occurrence of adverse events: Adverse events reported by subjects.
Tolerability and patient comfort | Visit 3 (Week 5), Visit 5 (Week 10)
  will be evaluated using a visual analog scale with a score from 0 to 10, with the latter representing the maximum comfort reported by the patient; measurements will be taken at the end of each of the study's scheduled sessions.
Degree of dyspnea | Visit 3 (Week 5), Visit 5 (Week 10)
  Will be assessed using the modified Medical Research Council (mMRC) scale from 0 to 4, with the latter representing the most severe degree of dyspnea. This measurment will be taken the end of each physiotherapy session scheduled in the study.
Volume of sputum (mL) | Visit 3 (Week 5), Visit 5 (Week 10)
  Recorded during the four weeks of treatment with each device using data reported in the "sputum diary"
Quality of Sputum | Visit 3 (Week 5), Visit 5 (Week 10)
  Measured according Murray sputum colour chart stratifies patients according to the presence of mucous (M), muco-purulent (MP) or purulent (P) sputum, during the four weeks of treatment with each device using data reported in the "sputum diary".
Number of exacerbations: Exacerbations reported by subjects. | Visit 3 (Week 5), Visit 5 (Week 10)
  Defined as a deterioration for at least 48 hours of three or more of the following key symptoms: cough, sputum volume or characteristics, sputum purulence, dyspnea and/or exercise intolerance, fatigue, malaise, and hemoptysis, associated with the clinician's belief that a change in treatment for bronchiectasis is necessary, occurring during the 4 weeks of treatment with each of the tested respiratory physiotherapy device
Quality of life | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  -Quality of life: will be assessed using the Quality-of-Life Bronchiectasis - QoL-B questionnaire
Health for bronchiectatic patients | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  -Health for bronchiectatic patients: measured using the Bronchiectasis Health Questionnaire - BHQ
Respiratory quality of life | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  -Respiratory quality of life: will be assessed using the Saint George Respiratory Questionnaire - SGRQ
Cough | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  -Cough: measured using the Leicester Cough Questionnaire - LCQ
Sleep Quality | V1 (Baseline), V3 (Week 5), V5 (Week 10)
  -Sleep quality: assessed using the Pittsburgh Sleep Quality Index. The global PSQI score ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Respiratory and Critical Care Unit, IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spinou A, Hererro-Cortina B, Aliberti S, Goeminne PC, Polverino E, Dimakou K, Haworth CS, Loebinger MR, De Soyza A, Vendrell M, Burgel PR, McDonnell M, Sutharsan S, Skrgat S, Maiz-Carro L, Sibila O, Stolz D, Kauppi P, Bossios A, Hill AT, Clifton I, Crichton ML, Walker P, Menendez R, Borekci S, Obradovic D, Nowinski A, Amorim A, Torres A, Lorent N, Welte T, Blasi F, Jankovic Makek M, Shteinberg M, Boersma W, Elborn JS, Chalmers JD, Ringshausen FC; EMBARC Registry Collaborators. Airway clearance management in people with bronchiectasis: data from the European Bronchiectasis Registry (EMBARC). Eur Respir J. 2024 Jun 6;63(6):2301689. doi: 10.1183/13993003.01689-2023. Print 2024 Jun. PMID 38609097